CLINICAL TRIAL: NCT02837614
Title: Evaluation of Preoperative Submucosal Dexamethasone in Third Molar Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qian Tao, Dr, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SunYat
Record Dates: First submitted 2016-06-25; First posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Impacted Third Molar Tooth
MeSH Terms: interventions — dexamethasone acetate; Amoxicillin; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (intramuscular dexamethasone) (Active Comparator): In Group A patients, 1 ml of dexamethasone (4mg) administered in the deltoid muscle before commencement of surgical procedure
  Interventions: Drug: dexamethasone acetate; Procedure: Third molar surgery
- Group B (submucosal dexamethasone) (Experimental): In Group B patients, 1 ml of dexamethasone was administered in submucosa after local anesthesia
  Interventions: Drug: submucosal dexamethasone injection; Procedure: Third molar surgery; Drug: Amoxicillin and paracetamol
- Group C (control) (Placebo Comparator): Group C patients continued without receiving any preoperative medication.
  Interventions: Procedure: Third molar surgery; Drug: Amoxicillin and paracetamol

INTERVENTIONS:
Drug: dexamethasone acetate — 1 milliliter of dexamethasone (4milligram) administered in the deltoid muscle before commencement of surgical procedure
  Arms: Group A (intramuscular dexamethasone)
Drug: submucosal dexamethasone injection — Local anesthesia was achieved using 2% lignocaine hydrochloride and 1:100 000 adrenaline and a standard technique was followed to block Inferior alveolar, lingual and long buccal nerve in all patients. In Group B patients, 1 ml of dexamethasone was administered in submucosa. Investigators divided 1 ml Dexamethasone is into 0.4 milliliter, 0.3 milliliter and 0.3 milliliter parts. Following the local anesthesia, each part of dexamethasone was injected submucosally in the buccal, lingual and retromolar region around the tooth to be extracted. Bone removal done around the tooth using a round bur under copious 0.9% normal saline irrigation and tooth elevated. The flap was sutured using three simple interrupted 3-0 black braided silk suture. All patients were given amoxicillin 500 milligram every 8 hours orally for 5 days, and 500 milligram of paracetamol postoperatively.
  Arms: Group B (submucosal dexamethasone)
Procedure: Third molar surgery — Surgical access was gained through standard Terrence Ward's incision to raise a full thickness mucoperiosteal flap. Bone removal done around the tooth using a round bur under copious 0.9% normal saline irrigation. The tooth sectioned at cemento-enamel junction whenever required and a Coupland elevator is used to elevate tooth or fragmented tooth out of socket. The socket examined for any debris and sharp bony margins smoothened. The empty socket was irrigated copiously and flap was sutured using three simple interrupted 3-0 black braided silk suture.
Drug: Amoxicillin and paracetamol — Amoxicillin 500 milligram every 8 hours orally for 5 days, and 500 milligram of paracetamol postoperatively (every 6 hours 1 tablet for 2 days).
  Arms: Group B (submucosal dexamethasone); Group C (control)

SUMMARY:
The study composed of sixty patients, each of whom required surgical extraction of a single impacted mandibular third molar under local anaesthesia. The patients were randomly allocated to one of 3 groups of 20 each. The three groups were categorized as Group A (intramuscular dexamethasone), Group B (submucosal dexamethasone) and Group C (control). The objective measurements of facial pain, swelling, and trismus was performed by an independent examiner at baseline (preoperatively), and at days 1, 3, and 7 postoperatively.

DETAILED DESCRIPTION:
The study was conducted as a prospective randomized comparative clinical study at the Department of Oral and Maxillofacial Surgery, Guanghua School of Stomatology, Sun Yat-sen University, Guangzhou and included 60 patients who needed surgical removal of a single impacted mandibular third molar under local anaesthesia. The study included 37 male and 13 female with age ranging from 20 to 40 years. Ethical approval was obtained from the Institutional Ethics Committee of Guanghua School of Stomatology, Sun Yat-sen University prior to the beginning of the study. The signed consent form obtained from all the patients after explaining the risks and benefits of the surgical procedure.

All the Sixty patients were randomly assigned to one of 3 groups of 20 each irrespective of age and sex using single-blind technique. The three groups were categorized as Group A (intramuscular dexamethasone), Group B (submucosal dexamethasone) and Group C (no steroid). Group A was given 8mg intramuscular dexamethasone, Group B was administered with 4mg submucosal dexamethasone and the Group C had no steroid injection.

The surgical procedure performed was same for all patients by the same operator. Local anesthesia was achieved using 2% lignocaine hydrochloride and 1:100 000 adrenaline and a standard technique was followed to block Inferior alveolar, lingual and long buccal nerve in all patients. In Group A patients, 1 ml of dexamethasone (4mg) administered in the deltoid muscle before commencement of surgical procedure. In Group B patients, 1 ml of dexamethasone was administered in submucosa after local anesthesia and the Group C patients continued without receiving any preoperative medication. In Group B, to standardize the drug delivery in third molar region the investigators followed the method described by Arakeri et al.6 for third molar surgery. According to the technique, the investigators divided 1 ml Dexamethasone (4mg) is into 0.4 ml, 0.3 ml and 0.3ml parts. Following the local anesthesia, each part of dexamethasone was injected submucosally in the buccal (0.3 ml), lingual (0.3 ml) and retromolar (0.4 ml) region around the tooth to be extracted (Figure1, 2, 3).

Surgical access was gained through standard Terrence Ward's incision to raise a full thickness mucoperiosteal flap. Bone removal done around the tooth using a round bur under copious 0.9% normal saline irrigation. The tooth sectioned at cemento-enamel junction whenever required and a Coupland elevator is used to elevate tooth or fragmented tooth out of socket. The socket examined for any debris and sharp bony margins smoothened. The empty socket was irrigated copiously and flap was sutured using three simple interrupted 3-0 black braided silk suture. A small gauze pack was placed over the wound and routine post-extraction instructions advised to patient. The duration of procedure from incision to the last suture was documented.

All patients were given amoxicillin 500 mg every 8 h orally for 5 days, and 500 mg of paracetamol postoperatively (every 6 h 1 tablet for 2 days). Patients are instructed to not to seek medical help for any postoperative discomfort without prior information to the surgeon.

The patients were recalled postoperatively on 1-, 3 and 5 days to record swelling, trismus and pain.

Pain, mouth opening, and facial swelling were objectively recorded at the first, third, and seventh postoperative days by an independent examiner.

Postoperative pain was assessed using a visual analog scale (VAS) of 10 point scale with a score of 0 measured "no pain" and 10 correspond to "very severe pain".18 Mouth opening was measured using the maximum distance between the maxillary central incisors and the mandibular central incisors. The difference between sum of post-operative measurements and sum of pre-operative measurements was considered as trismus. The evaluation of the facial swelling was performed by modification of Schultze-Mosgau et al method,19 and the facial measurements involved: 1. Tragus to the oral commissure 2.Tragus to the pogonion. The difference between sum of post-operative facial measurements and sum of pre-operative facial measurements was considered as facial swelling.

The data were tabulated and electronically stored. Descriptive statistics were mean (standard deviation) used to present the data. Chi square test and the analysis of variance (ANOVA), as appropriate, was used to assess the significance of differences. The level of significance less than 0.05 (P < 0.05) were considered as significant. Statistical analysis was performed using Statistical Package for the Social Sciences (SPSS) version 21

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) class I individuals
* Patients age between 18 - 40 years of age,
* Patients presenting with diagnosis of Class II position B impaction (Pell and Gregory classification)
* Patients who consent for regular recall visits

Exclusion Criteria:

* Patients having acute infection at extraction site
* Pregnant or lactating condition
* Smoking or tobacco/areca nut chewing habit
* Any systemic disease or medication therapy that could interfere with wound healing
* Impacted tooth associated with periapical infection or lesion
* Poor oral hygiene
* Patients with immunocompromise conditions

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Assessment of pain | 1 week
  Postoperative pain was assessed using a visual analog scale (VAS) of 10 point scale with a score of 0 measured "no pain" and 10 correspond to "very severe pain".
Trismus | 1 week
  Mouth opening was measured using the maximum distance between the maxillary central incisors and the mandibular central incisors. The difference between sum of post-operative measurements and sum of pre-operative measurements was considered as trismus.
Facial Swelling | 1 week
  The evaluation of the facial swelling was performed by modification of Schultze-Mosgau et al method, and the facial measurements involved: 1. Tragus to the oral commissure 2.Tragus to the pogonion. The difference between sum of post-operative facial measurements and sum of pre-operative facial measurements was considered as facial swelling.

IPD SHARING:
Plan to Share IPD: No